CLINICAL TRIAL: NCT05723822
Title: A Pilot Study to Explore the Effects of Lower-Leg Mechanical Tactile Sensory Stimulation on the Gait Speed of Mildly Cognitively Impaired Individuals
Brief Title: Effects of Walkasins on Gait Speed of Individuals With Mild Cognitive Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxFunction Inc. (Industry)
Collaborators: Innovative Design Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP 0007
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Cognitive Decline; Gait Disorders in Old Age
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Walkasins and PhySens-IMM System--Single Arm (Experimental): Participants who meet the eligibility criteria will don a pair of Walkasins and the PhySens-IMM System. They will perform some brief balance exercises (i.e., sensory integration exercises) and then complete the outcome assessments with their Walkasins turned off and without the use of an assistive device. After a rest period of about five minutes, they will repeat the outcome assessments with their Walkasins turned on.
  Interventions: Device: Walkasins

INTERVENTIONS:
Device: Walkasins — Walkasins is a non-invasive, wearable, lower limb sensory prosthesis, prescribed by a healthcare professional for long-term daily use as a prosthesis. It directly replaces the part of the function of the sensory end organs that persons with peripheral neuropathy have lost, the sensation in the soles of their feet. The system is comprised of two primary operating components:
  * A Receptor Sole, properly placed in the shoe, detects and transmits plantar pressure information normally performed by the mechanoreceptors and distal axons in the soles of the feet.
  * A Haptic Module, worn around the lower leg, generates directional specific mechanical tactile stimuli that produce action potentials that signal relevant balance information to the nervous system.

SUMMARY:
The primary aim of this pilot study is to investigate the effect of Walkasins, a wearable lower-limb sensory prosthesis, on the gait speed and balance function of participants with mild cognitive impairment as measured by the Saint Louis University Mental Status (SLUMS) Examination.

DETAILED DESCRIPTION:
The Walkasins system is one of a growing number of wearable devices that use various modalities of neuromodulation, defined as "the alteration of nerve activity through targeted delivery of a stimulus . . . to specific neurological sites in the body" (https://www.neuromodulation.com/). Because these technologies are relatively new, innovative applications of their use in various patient populations may lead to improvements in the care and quality of life of individuals who suffer from these life-altering diagnoses.

Previous studies of Walkasins have shown that individuals with peripheral neuropathy who have gait and balance problems walk faster with the Walkasins device. This increase may be related to an improved automaticity of gait function, which decreases the need for cognitive attention to the walking task, which is known to slow down gait. Individuals with mild cognitive impairment commonly show slow gait speeds, likely due to a decline in executive function. There is a reason to think that sensory stimuli from the Walkasins device can improve the automaticity of gait in these individuals and thereby enhance gait speed.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory person who is at least 65 years of age
* Ability to understand and provide informed consent
* Ability to perceive vibrations from the Walkasins Haptic Module
* Ability to complete the functional outcome measures without the use of an assistive device
* Foot size that allows the Walkasins to function appropriately
* Mild Cognitive Impairment (MCI) as measured by the Saint Louis University Mental Status (SLUMS) Exam (scores between 20 and 24 + or -2 for those with less than a high school education and scores between 21-26 + or -2 for those who graduated from high school, which indicate mild cognitive impairment) and/or a diagnosis of MCI (or related term) in the person's medical record
* Slow gait speed (<1m/second or slightly faster, provided all other criteria are met)

Exclusion Criteria:

* Use of ankle-foot orthosis for ambulation that prevents donning of Walkasins
* Self-reported acute thrombophlebitis including deep vein thrombosis
* Untreated lymphedema
* Untreated lesion of any kind, swelling, infection, inflamed area of skin or eruptions on the lower leg near product use
* Untreated fractures in the foot and ankle
* Self-reported severe peripheral vascular disease
* Other neurological conditions that impact walking (e.g., peripheral neuropathy)
* Weighs more than 300 pounds

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Condon, MSEE, Principal Investigator — Innovative Design Labs
Locations (1):
- The Pillars at Prospect Park, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oddsson LIE, Bisson T, Cohen HS, Iloputaife I, Jacobs L, Kung D, Lipsitz LA, Manor B, McCracken P, Rumsey Y, Wrisley DM, Koehler-McNicholas SR. Extended effects of a wearable sensory prosthesis on gait, balance function and falls after 26 weeks of use in persons with peripheral neuropathy and high fall risk-The walk2Wellness trial. Front Aging Neurosci. 2022 Sep 20;14:931048. doi: 10.3389/fnagi.2022.931048. eCollection 2022. PMID 36204554
- [Background] Koehler-McNicholas SR, Danzl L, Cataldo AY, Oddsson LIE. Neuromodulation to improve gait and balance function using a sensory neuroprosthesis in people who report insensate feet - A randomized control cross-over study. PLoS One. 2019 Apr 30;14(4):e0216212. doi: 10.1371/journal.pone.0216212. eCollection 2019. PMID 31039180
- See also: Walkasins Provider--RxFunction Company Website — https://www.rxfunction.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Walkasins and PhySens-IMM System--Single Arm: Participants who meet the eligibility criteria will don a pair of Walkasins and the PhySens-IMM System. They will perform some brief balance exercises (i.e., sensory integration exercises) and then complete the outcome assessments first with their Walkasins turned off and without the use of an assistive device. After a rest period of about five minutes, they will repeat the outcome assessments with their Walkasins turned on.
Period: Overall Study
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 84.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Saint Louis University Mental Status (SLUMS) Test [Mean (Standard Deviation); unit: Score on a Scale] — The Saint Louis University Mental Status (SLUMS) test is an assessment tool for dementia and mild cognitive impairment. It consists of 11 items with a minimum score of 0 and a maximum score of 30. For those with less than a high school education, scores of 25-30 indicate normal cognition; scores of 20-24 indicate mild neurocognitive disorder; and scores of 1-19 indicate dementia. For those with a high school education, scores of 27-30 indicate normal cognition; scores of 21-26 indicate mild neurocognitive disorder; and scores of 1-20 indicate dementia.
  Score on a Scale | 23.5 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in 4-Meter Gait Speed (Section 2 of the Short Physical Performance Battery)
Description: The 4-meter gait speed test measures the number of seconds it takes a person to walk four meters on a level surface. Gait speed measures are a significant indicator of a person's functional mobility. Higher gait speeds (meters/second) are better than lower gait speeds and are indicative of better functional mobility. (Generally, gait speeds less than 1m/second are considered slow.)
Time Frame: 3 Times During 1 Session <1.5 Hours (Screening + Walkasins Off Condition then Walkasins On Condition)
Measure: Mean (Standard Deviation); unit: Meters/Second
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Number analyzed (Participants) | 12
Meters/Second
  Baseline Assessment for Eligibility | 0.79 (0.16)
  Walkasins OFF | 0.82 (0.18)
  Walkasins ON | 0.79 (0.20)

2. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery measures walking speed, standing balance, and sit-to-stand performance. Scores on balance, gait speed, and chair-stand tests are added (summed) for a total score. (Scores on balance, gait speed, and chair-stand tests are not reported separately since they are not "subscales" per se.) SPPB scores may range from 0 to 12. Higher total scores indicate better balance and gait.
Time Frame: Twice During 1 Session <1.5 Hours (Walkasins Off Condition then Walkasins On Condition)
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Single Arm: Participants who meet all eligibility criteria will don a pair of Walkasins and the PhySens-IMM System. They will perform some brief balance exercises (i.e., sensory integration exercises) and then complete the outcome assessments first with their Walkasins turned off and without the use of an assistive device. After a brief rest period, they will repeat the outcome assessments with their Walkasins turned on.
  Walkasins: The Walkasins System is a prosthetic device that replaces part of the function of the nerves in the feet that are used to detect and inform the brain about foot contact with the ground, which is critical for maintaining balance during standing and walking activities. It provides directional mechanical tactile stimuli to the front, back, left, and right surfaces of the user's legs, relaying balance information to a location above the ankle where skin sensation is still present.
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Score on a Scale
  Walkasins OFF | 8.2 (1.9)
  .Walkasins ON | 7.5 (2.1)

3. Secondary Outcome: Timed Up and Go (TUG)
Description: The Timed Up and Go Test is part of the Centers for Disease Control (CDC)-recommended STEADI test protocol for balance function. From a seated position in a standard armchair, the participant is asked to stand up from the chair, walk to a line on the floor 10 feet away at normal pace, turn, walk back to the chair at normal pace, and sit down again. The tester records the time taken from the command "Go" until the subject sits down again. Lower times indicate better/faster performance.
Time Frame: Twice During 1 Session <1.5 Hours (Walkasins Off Condition then Walkasins On Condition)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Number analyzed (Participants) | 12
Seconds
  Walkasins OFF | 15.46 (5.4)
  Walkasins ON | 15.83 (5.66)

4. Secondary Outcome: Timed Up and Go Cognitive (TUG-COG)
Description: The TUG-COG is performed similarly to the TUG; however, the participant is also asked to count backwards by 3 from a randomly selected number between 20 and 100 while performing the TUG (standing up from the chair, walking to a line on the floor 10 feet away, turning, walking back to the chair at a normal pace, and sitting down again). Lower times indicate better/faster performance.
Time Frame: Twice During 1 Session <1.5 Hours (Walkasins Off Condition then Walkasins On Condition)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Number analyzed (Participants) | 12
Seconds
  Walkasins OFF | 21.64 (7.10)
  Walkasins ON | 18.85 (6.96)

5. Secondary Outcome: Falls Efficacy Scale
Description: The Falls Efficacy Scale is a 16-item questionnaire that measures an individual's fear of falling or concerns about falling during activities of daily living. Scores may range from 16 (not at all concerned) to 64 (very concerned). Lower scores are better than higher scores because they indicate less concern about falling.
Time Frame: Once During 1 Session <1.5 Hours
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
Number analyzed (Participants) | 12
Score on a Scale | 32.2 (7.6)

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored during the subject visits (lasting approximately 1.5 hours). No adverse events occurred during the study's duration.
Groups:
- Walkasins and PhySens-IMM System--Single Arm: Participants who meet the eligibility criteria will don a pair of Walkasins and the PhySens-IMM System. They will perform some brief balance exercises (i.e., sensory integration exercises) and then complete the outcome assessments first with their Walkasins turned off and without the use of an assistive device. After a brief rest period, they will repeat the outcome assessments with their Walkasins turned on.
Arm/Group | Walkasins and PhySens-IMM System--Single Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
This trial was an exploratory pilot study only, and as such, participants were not randomized. In addition, 75% of the participants were females, and only 12 individuals participated in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05723822/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT05723822/ICF_001.pdf